CLINICAL TRIAL: NCT04876521
Title: Comparative Efficacy and Safety of Low Dose Amisulpride Vs Olanzapine-Fluoxetine Combination in the Treatment of Post Schizophrenic Depression: A Randomized Controlled Trial
Brief Title: Low Dose Amisulpride Vs Olanzapine-Fluoxetine Combination in Post-Schizophrenic Depression
Acronym: PSD-AOFC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: All India Institute of Medical Sciences, Bhubaneswar (Other)
Responsible Party: Principal Investigator, BISWA RANJAN MISHRA, Additional Professor, Department of Psychiatry, All India Institute of Medical Sciences, Bhubaneswar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AIIMS BBSR/PGThesis/2019-21
Record Dates: First submitted 2021-05-03; First posted 2021-05-06 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Post-Schizophrenic Depression
Keywords: Post-Schizophrenic Depression; Amisulpride; Olanzapine-Fluoxetine Combination; Post Psychotic Depression
MeSH Terms: interventions — Amisulpride; olanzapine-fluoxetine combination

STUDY DESIGN:
Intervention Model Description: Randomized, parallel-group, rater-blinded, clinical trial.
Who Masked: Outcomes Assessor
Masking Description: The proposed study will be rater-blinded. The ratings would be done by a psychiatrist who would be blinded to the nature of the intervention provided
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amisulpride Group (Experimental): The patients will receive low dose Amisulpride at 100-300 mg/day.
  Interventions: Drug: Amisulpride
- Olanzapine-Fluoxetine Group (Active Comparator): the patients will receive Olanzapine-Fluoxetine Combinations at 5/10 + 20 mg/day.
  Interventions: Drug: Olanzapine-Fluoxetine Combination

INTERVENTIONS:
Drug: Amisulpride — low dose of Amisulpride at 100-300 mg/day
  Other Names: Sulpitac; Amazeo; Soltus
  Arms: Amisulpride Group
Drug: Olanzapine-Fluoxetine Combination — Olanzapine (5-10 mg/day) and Fluoxetine (20 mg/day)
  Other Names: Oleanz Fort; Oleanz Plus
  Arms: Olanzapine-Fluoxetine Group

SUMMARY:
Post-Schizophrenic Depression (PSD) increases the morbidity and mortality of Schizophrenic patients. Hence, it warrants early assessment and intervention. But, clinical trials on PSD are very few. However, an Antipsychotic with an adjunctive Antidepressant (like Olanzapine-Fluoxetine Combination) is the commonly prescribed treatment in PSD. Low dose Amisulpride (<400 mg/day) which is effective against the negative symptoms of Schizophrenia has also proved efficacious in treating depression in non-psychotic conditions, but its antidepressant property has never been studied in PSD. This is an 8-week, randomized, parallel-group study that will explore the efficacy and safety of low-dose Amisulpride versus Olanzapine-Fluoxetine Combination in the treatment of PSD. Our hypothesis is that low dose Amisulpride has better efficacy and safety versus Olanzapine-Fluoxetine Combination in PSD, after 8-weeks.

DETAILED DESCRIPTION:
The proposed study would be an 8-week, randomized, controlled, parallel-group, clinical trial which will be conducted at the Inpatient and Outpatient settings of the Department of Psychiatry, AIIMS, Bhubaneswar. Patients with the diagnosis of Post Schizophrenic Depression according to the ICD 10 (DCR) and meeting all the Inclusion and Exclusion Criteria would be selected for the study. At first, the patients and their family members/ guardians would be explained about the study procedure along with its possible risks and benefits using a Patient Information Sheet (in their local language). After obtaining a written Informed Consent from the Legally Authorised Relative, the patients would be finally recruited for the study.

All recruited patients would be randomized using computer-generated random numbers into two treatment groups with an allocation ratio of 1:1. The sociodemographic and clinical data of the patients would be collected as per the designed sheets. Then at baseline, the CDSS and CGI ratings would be assessed, and the serum BDNF would be tested for each patient. The study would be rater-blinded. The experimental group would receive Amisulpride at a low dosage of 100-300 mg/day and the control group would receive a combination of Olanzapine at 5mg or 10 mg/day and Fluoxetine at 20mg/day.

The two groups would be followed for 8 weeks, at the completion of which all the patients would be reassessed. The follow-up assessment would involve a re-evaluation of the CDSS and the CGI scores and the Serum BDNF levels to see for any change. The data thus collected would be analyzed, compared within and in between the study groups and statistical tests would be applied for drawing conclusions. The missing values will be analyzed by an intention-to-treat protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Post Schizophrenic Depression according to ICD10-DCR (International Classification of Diseases 10- Diagnostic Criteria for Research).
2. Aged between 18 to 60 years of either sex
3. Patients with a positive score of less than 29 on the Positive and Negative Syndrome Scale (PANSS) [88]
4. Patients with a score of more than 6 on the Montgomery-Asberg Depression Rating Scale (MADRS) [89-90]
5. Patients without Extrapyramidal symptoms: a score of less than 3 on the Simpson-Angus Scale [91]
6. With Informed consent from the Legally Authorised Relative

Exclusion Criteria:

1. Patients with a medical or neurological disorder
2. Patients with a history of substance dependence
3. Patients with high suicidality
4. Patients with a past history of primary depression
5. Patients already on Olanzapine-Fluoxetine combination or Amisulpride

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2021-06-09 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Biswa R Mishra, MD, Principal Investigator — All India Institute of Medical Sciences, Bhubaneswar
Locations (1):
- All India Institute of Medical Sciences, Bhubaneswar, Odisha, India

IPD SHARING:
Plan to Share IPD: No
To maintain the confidentiality of the participants.

REFERENCES:
- [Background] Berrios GE, Bulbena A. Post psychotic depression: the Fulbourn cohort. Acta Psychiatr Scand. 1987 Jul;76(1):89-93. doi: 10.1111/j.1600-0447.1987.tb02866.x. PMID 3630758
- [Background] Stern MJ, Pillsbury JA, Sonnenberg SM. Postpsychotic depression in schizophrenics. Compr Psychiatry. 1972 Nov-Dec;13(6):591-8. doi: 10.1016/0010-440x(72)90060-0. No abstract available. PMID 4637572
- [Background] Rahim T, Rashid R. Comparison of depression symptoms between primary depression and secondary-to-schizophrenia depression. Int J Psychiatry Clin Pract. 2017 Nov;21(4):314-317. doi: 10.1080/13651501.2017.1324036. Epub 2017 May 15. PMID 28503978
- [Background] Whitehead C, Moss S, Cardno A, Lewis G. Antidepressants for the treatment of depression in people with schizophrenia: a systematic review. Psychol Med. 2003 May;33(4):589-99. doi: 10.1017/s0033291703007645. PMID 12785461
- [Background] Addington D, Addington J, Schissel B. A depression rating scale for schizophrenics. Schizophr Res. 1990 Jul-Aug;3(4):247-51. doi: 10.1016/0920-9964(90)90005-r. PMID 2278986
- [Background] Moller HJ. Amisulpride: limbic specificity and the mechanism of antipsychotic atypicality. Prog Neuropsychopharmacol Biol Psychiatry. 2003 Oct;27(7):1101-11. doi: 10.1016/j.pnpbp.2003.09.006. PMID 14642970
- [Background] Bocchio-Chiavetto L, Bagnardi V, Zanardini R, Molteni R, Nielsen MG, Placentino A, Giovannini C, Rillosi L, Ventriglia M, Riva MA, Gennarelli M. Serum and plasma BDNF levels in major depression: a replication study and meta-analyses. World J Biol Psychiatry. 2010 Sep;11(6):763-73. doi: 10.3109/15622971003611319. PMID 20334574
- [Derived] Biswas T, Mishra BR, Maiti R, Padhy SK, Mishra A. Efficacy and safety of low-dose amisulpride versus olanzapine-fluoxetine combination in post-schizophrenic depression: A randomized controlled trial. J Psychiatr Res. 2024 May;173:302-308. doi: 10.1016/j.jpsychires.2024.03.048. Epub 2024 Mar 28. PMID 38560960

RESULTS

PARTICIPANT FLOW:
Groups:
- Amisulpride Group: The patients received Amisulpride at 100-300 mg/day.
  Amisulpride: Amisulpride at 100-300 mg/day
- Olanzapine-Fluoxetine Group: the patients received Olanzapine-Fluoxetine Combinations at 5/10-5/20 mg/day.
  Olanzapine-Fluoxetine Combination: Olanzapine (5 mg/day) and Fluoxetine (10-20 mg/day)
Period: Overall Study
Arm/Group | Amisulpride Group | Olanzapine-Fluoxetine Group
Started | 30 | 30
Completed | 25 | 23
Not Completed | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Amisulpride Group: Received Amisulpride at 100-300 mg/day
- Olanzapine-Fluoxetine Group: Received Olanzapine-Fluoxetine Combination: Olanzapine (5-10 mg/day) and Fluoxetine (20 mg/day)
- Total: Total of all reporting groups
Arm/Group | Amisulpride Group | Olanzapine-Fluoxetine Group | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.2 (10.1) | 35.4 (9.8) | 35.3 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 17 | 18 | 35
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
PANSS-P score [Mean (Standard Deviation); unit: score on a scale] — The Positive and Negative Syndrome Scale - Positive (PANSS-P) is a medical scale that measures the severity of positive symptoms of schizophrenia. It has seven items (delusions, conceptual disorganization, hallucinations, excitement, grandiosity, suspiciousness/persecution and hostility). Each item has a score range of 1 to 7. Thus, the total minimum score is 7, and the total maximum score is 49. Higher scores mean more severity of symptoms.
  score on a scale | 13.70 (4.44) | 13.80 (4.22) | 13.75 (4.29)
MADRS score [Mean (Standard Deviation); unit: score on a scale] — The Montgomery-Asberg Depression Rating Scale (MADRS) is a ten-item scale used to measure the severity of depressive symptoms in a patient. Each item has a score ranging from 0 to 6. Thus, the total minimum score is 0, and the total maximum score is 60. The higher the score, the more severe the depressive symptoms.
  score on a scale | 23.17 (6.49) | 23.73 (6.82) | 23.45 (6.61)

OUTCOME MEASURES:

1. Primary Outcome: Calgary Depression Scale for Schizophrenia (CDSS)
Description: Calgary Depression Scale for Schizophrenia (CDSS) scores is used to measure the severity of depressive symptoms in the study groups. The total score ranges from 0 - 36. Higher scores represent a higher severity of depression.
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Amisulpride Group | Olanzapine-Fluoxetine Group
Number analyzed (Participants) | 25 | 23
score on a scale | 8.31 (0.47) | 8.62 (0.60)

2. Secondary Outcome: Clinical Global Impression - Severity (CGI) Scale
Description: The Clinical Global Impression - Severity (CGI-S) is a 7-point scale used to measure the severity of the illness in the study groups [minimum: 1 and maximum 7]: Higher scores mean higher severity of disease.
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Amisulpride Group | Olanzapine-Fluoxetine Group
Number analyzed (Participants) | 25 | 23
units on a scale | 3.31 (0.09) | 3.44 (0.11)

3. Secondary Outcome: Serum BDNF Levels
Description: The change in serum BDNF levels in the study groups at 8 weeks (in pg/mL)
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: picograms per milliliter
Arm/Group | Amisulpride Group | Olanzapine-Fluoxetine Group
Number analyzed (Participants) | 25 | 23
picograms per milliliter | 1453.59 (44.62) | 1471.19 (48.22)

4. Secondary Outcome: Correlation
Description: Determine the correlation (if any) between the changes in CDSS scores and serum BDNF levels. The correlation coefficient is represented as r, with values from -1 to +1 [where +/- 1 mean strongest correlation and 0 mean no correlation].
Time Frame: 8 week
Measure: Number; unit: r (correlation coefficient)
Arm/Group | Amisulpride Group | Olanzapine-Fluoxetine Group
Number analyzed (Participants) | 25 | 23
r (correlation coefficient) | -0.161 | -0.123

5. Secondary Outcome: Adverse Drug Reactions
Description: Detect adverse drug reactions (if any) and grading their severity
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Amisulpride Group | Olanzapine-Fluoxetine Group
Number analyzed (Participants) | 25 | 23
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Amisulpride Group | Olanzapine-Fluoxetine Group
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

LIMITATIONS AND CAVEATS:
1. Small sample size
2. Single-center study
3. No control arm for comparing the Serum BDNF levels

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-06-01): https://cdn.clinicaltrials.gov/large-docs/21/NCT04876521/Prot_SAP_ICF_000.pdf